CLINICAL TRIAL: NCT01201590
Title: The Effects of Cocoa Flavanols on Insulin Resistance in at 'At-risk' Population
Brief Title: The Effects of Cocoa Flavanols on Insulin Resistance in an 'At-risk' Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1000165377
Record Dates: First submitted 2009-09-30; First posted 2010-09-14 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; obesity; cocoa; women
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flavanol Cocoa (Experimental): 609mg cocoa flavanols per 24g serving
  Interventions: Dietary Supplement: High Flavanol Cocoa
- Low flavanol cocoa (Placebo Comparator): 13mg cocoa flavanols per 24g serving
  Interventions: Dietary Supplement: Low Flavanol Cocoa

INTERVENTIONS:
Dietary Supplement: High Flavanol Cocoa — cocoa consumed as a 24g dairy based cocoa drink mix, twice a day (mid-morning & early evening on an empty stomach), for 4 weeks.
  Arms: High Flavanol Cocoa
Dietary Supplement: Low Flavanol Cocoa — cocoa consumed as a 24g dairy based cocoa drink mix, twice a day (mid-morning & early evening on an empty stomach), for 4 weeks.
  Arms: Low flavanol cocoa

SUMMARY:
The aim of the current study is to investigate the ability of antioxidants found in cocoa ('flavanols') to increase the body's sensitivity to the hormone insulin. 32 overweight or mildly obese women, who are otherwise healthy, will be recruited. Subjects will attend the laboratory on 3 occasions after fasting from midnight. The 1st visit is a medical screening, with laboratory visits 2 and 3 separated by 4 weeks, during which time subjects will consume a cocoa drink (containing either high or low amounts of flavanols) twice a day. Subjects will record their food intake for 3-days before visit 2 and in week 3 of consuming the cocoa. They will also eat a diet of standard macronutrient composition for 3 days before visits 2 and 3. During the 5 hour laboratory visits, subjects will have a scan to assess their body composition using a low-dose x-ray machine (Dual Energy X-ray Absorptiometry; DEXA), and have their insulin sensitivity measured using a 3 hour hyperinsulinemic, euglycaemic Clamp.

DETAILED DESCRIPTION:
Background; Overweight and mild obesity are associated with insulin resistance and mild elevations in lipid risk factors which are not usually sufficiently abnormal to merit treatment. Such people are encouraged to lose weight to reduce their risk of progressing to type 2 diabetes and coronary heart disease, but there is clearly a potential role for dietary modifications to maximize any potential benefit of this weight loss. Cocoa flavanols (CF) are known to have vascular effects which might enhance substrate delivery to metabolically active tissues, and thus improve insulin sensitivity.

Aims; This randomized, double blind, placebo controlled, parallel design study aims to investigate the longer term effects of CF intake on insulin sensitivity. It is hypothesized that studying otherwise healthy overweight and mildly obese subjects, with evidence of fasting insulin resistance, would show whether there was potential benefit of CF in an 'at risk' population.

Experimental protocol and methods; 32 overweight or obese women (Body Mass Index 27-35), who are otherwise healthy, will be recruited onto the study. They will attend the 'David Greenfield Human Physiology' laboratories on 3 convenient mornings, following an overnight fast. The 1st visit is a medical screening and will involve signing a consent form, completing a medical screening and food frequency questionnaire, having height, weight, hip/waist circumference measurements taken and a 10ml sample of blood taken for routine analysis. Subjects will then be asked to complete a 3-day diet diary for macronutrient assessment and to consume a diet providing 50% of energy as carbohydrate for 3 days prior to the 2nd laboratory visit. This 2nd visit will involve having a DEXA body composition scan and a 3-hour hyperinsulinaemic, euglycaemic glucose clamp. Starting on the following morning, subjects will then consume a cocoa drink (containing either 450mg or 25mg of CF) twice a day for 28 days. A 3-day diet diary for macronutrient assessment will be recorded during week 3 of taking the cocoa and a standardized diet will be consumed for 3 days prior to the final laboratory visit, as before. This 3rd visit will be identical to visit 2 and occur immediately after 28days of taking the cocoa.

Measurable end points Insulin sensitivity 'M' value (mg glucose disposal from the blood/kg body weight.min), Respiratory exchange ratio, Resting metabolic rate, Homeostatic model assessment for insulin resistance (HOMA-IR) Body composition (DEXA) Macronutrient composition of the diet before and during the intervention period

ELIGIBILITY:
Inclusion Criteria:

* female,
* aged > 18 years,
* pre-menopausal,
* Body Mass Index (BMI)27-35,
* homeostatic model assessment-Insulin Resistance(HOMA-IR)value > 1.5,
* daily consumption of caffeine containing foods/drinks

Exclusion Criteria:

* pregnant or breast feeding,
* any metabolic or endocrine abnormalities,
* clinically significant abnormalities on screening,
* fasting glucose > 6.0mmol/l,
* taking medication other than the contraceptive pill,
* herbal supplement use,
* food allergies related to the investigational product (cocoa, peanuts, milk)
* sensitivity to methylxanthines (e.g., caffeine, theobromine)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in Insulin sensitivity 'M' value (mg glucose disposal from the blood/kg body weight/min), | after 28 days of supplementation
  Insulin sensitivity calculated from glucose disposal during a hyperinsulinemic, euglycemic glucose clamp

SECONDARY OUTCOMES:
Change in Glucose Oxidation rate | after 28 days of supplementation
  Measured by ventilated hood indirect calorimetry during the glucose clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Physiology Laboratories, University of Nottingham, Nottingham, Notts, United Kingdom

REFERENCES:
- [Result] Simpson EJ, Mendis B, Dunlop M, Schroeter H, Kwik-Uribe C, Macdonald IA. Cocoa Flavanol Supplementation and the Effect on Insulin Resistance in Females Who Are Overweight or Obese: A Randomized, Placebo-Controlled Trial. Nutrients. 2023 Jan 21;15(3):565. doi: 10.3390/nu15030565. PMID 36771271